CLINICAL TRIAL: NCT00018941
Title: Phase III Randomized Study of Intravenous Low Dose Versus Intravenous High Dose Versus Subcutaneous Interleukin-2 for Metastatic Renal Cell Carcinoma
Brief Title: Interleukin-2 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000076799; NCI-91-C-0094; NCI-T91-0053N; NCT00001268 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-05-05 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2003-03

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. It is not yet known which regimen of interleukin-2 is most effective for kidney cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of different regimens of interleukin-2 in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and overall survival of patients with metastatic renal cell carcinoma treated with either low-dose or high-dose intravenous interleukin-2 (IL-2) or subcutaneous IL-2. II. Compare the toxic effects of these 3 regimens in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to presence of renal tumor (yes vs no). Patients are randomized to one of three treatment arms. Arm I: Patients receive low dose interleukin-2 (IL-2) IV every 8 hours for up to 15 doses. Treatment repeats in 7-10 days for one complete course. Arm II: Patients receive high dose IL-2 IV every 8 hours for up to 15 doses. Treatment repeats in 7-10 days for one complete course. Arm III: Patients receive IL-2 subcutaneously daily 5 days a week for 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease receive an additional complete course of therapy.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven, metastatic renal cell carcinoma with measurable disease No more than 25% of liver replaced with tumor No CNS involvement or major nerve compression allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: More than 3 months Hematopoietic: Not specified Hepatic: Bilirubin less than 2.0 mg/dL AST and ALT no greater than 3 times normal Renal: Creatinine less than 1.6 mg/dL Cardiovascular: Normal EKG Normal thallium stress test (required of patients 50 years of age and older or as clinically indicated) Pulmonary: FEV1 and VC greater than 65% of predicted (pulmonary function screening required of patients with significant smoking history or suspicion of pulmonary disease) Other: No second malignancy, except: Basal cell skin cancer Carcinoma in situ of the cervix No significant psychiatric disease that would preclude consent or treatment No systemic infection No coagulation disorders or bleeding Not pregnant HIV negative

PRIOR CONCURRENT THERAPY: No prior therapy within 28 days Biologic therapy: No prior interleukin-2 Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No concurrent steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1991-04; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Yang, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States

REFERENCES:
- [Result] Yang JC, Topalian SL, Parkinson D, Schwartzentruber DJ, Weber JS, Ettinghausen SE, White DE, Steinberg SM, Cole DJ, Kim HI, et al. Randomized comparison of high-dose and low-dose intravenous interleukin-2 for the therapy of metastatic renal cell carcinoma: an interim report. J Clin Oncol. 1994 Aug;12(8):1572-6. doi: 10.1200/JCO.1994.12.8.1572. PMID 8040669